CLINICAL TRIAL: NCT01319435
Title: Phase I, Open-label Study to Evaluate the Pharmacokinetics and Tolerability of Ciprofloxacin in Neonates With Suspected or Proven Gram Negative Infection
Brief Title: TINN Pharmacokinetics (PK) Study Treat Infections iN Neonates
Acronym: TINN-PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LWH0852; 2010-019955-23 (EudraCT Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Pharmacokinetics of Ciprofloxacin in Neonates
Keywords: Ciprofloxacin; Neonates; Gram negative infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacokinetics of ciprofloxacin (Other): Patients receiving ciprofloxacin following clinical decision by attending physician
  Interventions: Procedure: Collection of biological samples

INTERVENTIONS:
Procedure: Collection of biological samples — Sparse blood samples (n=2 or 3 depending on weight) will be drawn on day 1 and day 5- 7 (or last day of treatment if the course is completed before day 7).
  Monitoring of adverse events DNA for pharmacogenetics (scavenged clinical samples or buccal) CSF (if required clinically) Faeces

SUMMARY:
Phase I, open-label study to evaluate the pharmacokinetics, tolerability and short-term safety of ciprofloxacin in neonates with suspected (or proven) Gram Negative infection. Objectives: To evaluate the multiple-dose pharmacokinetics of ciprofloxacin in neonates and young infants (24 - 52 weeks postmenstrual age) with suspected or proven Gram Negative infection.

To evaluate the tolerability and describe short-term safety of ciprofloxacin in neonates and young infants with suspected (or proven) Gram Negative infection.

To describe the clinical outcomes of neonates treated with ciprofloxacin

DETAILED DESCRIPTION:
This study is part of TINN 'Treat Infections in Neonates' a comprehensive project that is evaluating the safety of ciprofloxacin and how it is tolerated by neonates. Ciprofloxacin is an antibiotic that has been used for many years in newborn babies and infants less than 3 months old to treat bacteria that are resistant to other antibiotics. Ciprofloxacin is unlicensed for this age group. The European Medicines Agency and WHO have prioritised research about this drug. The TINN consortium aims to conduct the work required for a license (marketing authorization) in newborn babies and infants less than 3 months old. The aim of this study is to describe how newborn babies and young infants deal with this medicine. Blood samples will be taken at the beginning of the course of antibiotics and at the end. A minimal amount of blood will be required (less than half a teaspoon) in total and collected by staff experienced in blood sampling from neonates in a way that causes the least disruption to the baby. The levels of ciprofloxacin in the blood will be measured. The levels will be used to work out how quickly the body gets rid of the medicine. This will allow recommendations about the best dose and how often the medicine should be given.

We aim to recruit 50 neonates and infants under the age of 3 months who have been prescribed Ciprofloxacin as inpatients for suspected or proven infection. They will be recruited over 2 years from the neonatal unit at Liverpool Women's NHS Foundation Trust and Alder Hey Children's NHS Foundation Trust. Consent will be requested for babies to have more detailed investigation to see if there if genetic factors affect the way the body handles ciprofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ciprofloxacin following clinical decision by attending physician

Exclusion Criteria:

* Likely not to survive 48 hours in the judgement of attending physician
* Ciprofloxacin commenced before 5th day of life

Ages: 24 Weeks to 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Ciprofloxacin plasma concentration and population pharmacokinetic (PK) parameters | 6 weeks
  Ciprofloxacin plasma concentration and population pharmacokinetic (PK) parameters [maximum concentration, clearance, area under the curve (0-tau)], their relationship with selected covariates their interindividual variability (CV%). Covariate analysis will include postmenstrual age, gestational age, postnatal age, weight, and serum creatinine

SECONDARY OUTCOMES:
PK variables | 6 weeks
  PK variables, including apparent volume of distribution and half life.
Tolerability | 6 weeks
  Withdrawal due to lack of tolerability
Safety | 6 Weeks
  Adverse events (AEs) and serious adverse events (SAEs).
Clinical/microbiological outcomes | 6 Weeks
  Outcome of treatment episodes (clinical and microbiological)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Turner, MD, Principal Investigator — University of Liverpool/Liverpool Women's Hospital
Locations (2):
- United Kingdom (2):
  - Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside
  - Liverpool Women's NHS Foundation Trust, Liverpool, Merseyside